CLINICAL TRIAL: NCT01030081
Title: A Randomized Controlled Phase Ⅳ Trial With Two Equally Sized Treatment Groups: Amlodipine And Nifedipine GITS
Brief Title: Amlodipine Prevents Morning Blood Pressure Surge Study
Acronym: ARMORS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Ji-Guang Wang, Director, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ARMORS
Record Dates: First submitted 2009-12-10; First posted 2009-12-11 (Estimated); Last update posted 2014-05-22 (Estimated); Status verified 2014-05

CONDITIONS: Hypertension
Keywords: 24 hour blood pressure; morning blood pressure surge; amlodipine; nifedipine GITS
MeSH Terms: conditions — Hypertension | interventions — Amlodipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Amlodipine (Norvasc®) (Experimental)
  Interventions: Drug: Amlodipine (Norvasc®)
- Nifedipine GITS (Adalat® XL 30) (Active Comparator)
  Interventions: Drug: Nifedipine GITS (Adalat® XL 30

INTERVENTIONS:
Drug: Amlodipine (Norvasc®) — Amlodipine (Norvasc®), tablet, 5 mg
  Arms: Amlodipine (Norvasc®)
Drug: Nifedipine GITS (Adalat® XL 30 — Nifedipine GITS (Adalat® XL 30), controlled released tablet, 30 mg
  Arms: Nifedipine GITS (Adalat® XL 30)

SUMMARY:
1. Study name:Amlodipine Prevents Morning Blood Pressure Surge Study
2. Study drugs:amlodipine (Norvasc®) and nifedipine GITS (Adalat®)
3. Rationale: Several recent studies compared 24-h blood pressure lowering effect of these 2 dihydropyridine drugs, amlodipine and nifedipine GITS, but produced inconsistent results. Therefore, a randomized controlled trial with a larger sample size is required to compare these 2 dihydropyridines in the blood pressure control over 24 hours in general and during early morning hours and at night in particular.
4. Objective: The primary objective of this study is to test the hypothesis that amlodipine compared with nifedipine GITS has a stronger effect in preventing morning blood pressure surge (4 am to 8 am) in mild to moderate hypertensive patients.The secondary objective of the study is to compare the effects of amlodipine and nifedipine GITS in reducing nighttime blood pressure (10 pm to 4 am) in patients with a decreased nocturnal blood pressure fall.
5. Study design: The present study is designed as a randomized, actively controlled, multi-centre parallel group trial (phase Ⅳ) with two equally sized treatment groups: amlodipine and nifedipine GITS.
6. Study population: 500 hypertensive patients meet the inclusion/exclusion criteria.
7. Randomization and treatment: After stratification for centre, 500 eligible patients will be randomized into 2 groups. 250 will receive amlodipine 5 mg per day, and 250 will receive nifedipine GITS 30 mg per day. At 4 weeks of follow-up, the drug dosage per day may increase to 10 mg of amlodipine and 60 mg of nifedipine GITS, if blood pressure measured in doctor's office cannot be controlled to a level below 140/90 mm Hg. If there were no compelling indication, no other antihypertensive drug is allowed during the 2-month trial.
8. Follow up: All patients should give written informed consent at entry into the present study. In addition to 24-h ambulatory blood pressure monitoring, patients should also undergo a questionnaire survey and clinical measurements including clinic blood pressure. Patients will be followed up at the end of 4 weeks and 8 weeks after randomization.
9. Sample size estimation: The number of required subject for the whole trial is 500.
10. Timeline: October 2009 to July 2013.
11. Organization: The Centre for Epidemiological Studies and Clinical Trials, Ruijin Hospital, Shanghai, China.

DETAILED DESCRIPTION:
1. Study name: Amlodipine Prevents Morning Blood Pressure Surge Study (ARMORS)
2. Study drugs: amlodipine (Norvasc®) and nifedipine GITS (Adalat®)
3. Rationale:

Previous meta-analyses of randomized controlled trials have demonstrated that the long acting dihydropyridine calcium channel blocker amlodipine (Norvasc®), compared with other antihypertensive drugs, provides more protection against stroke. The benefit of amlodipine against stroke is approximately 10% greater than diuretics/β-blockers, and 20% greater than angiotensin-converting enzyme inhibitors and angiotensin receptor blockers. Of all the dihydropyridine calcium channel blockers, only amlodipine provides protection against myocardial infarction similar as angiotensin-converting enzyme inhibitors, diuretics and β-blockers, and more than angiotensin receptor blockers. The benefit of amlodipine in the prevention of stroke might be attributable to its 24-h blood pressure control.

24-h ambulatory blood pressure is more predictive of cardiovascular events than clinic pressure measured in doctor's office. The smoother the 24-h ambulatory blood pressure control, the lower the risk of target organ damage. Both systolic and diastolic blood pressure show a circadian rhythm with a nocturnal blood pressure fall and a morning blood pressure surge. The incidence of cardiovascular complications of hypertension, such as myocardial infarction and stroke, is higher in the early morning hours than the rest of the day. Several previous studies have demonstrated that an exaggerated morning blood pressure surge is associated with the incidence of stoke and with cardiovascular structural remodeling. Moreover, non-dipping of blood pressure at night (non-dipper, nighttime blood pressure fall less than 10%) is prevalent and is associated with a higher risk of cardiovascular event. In a recent study of controlled hypertensive patients, the prevalence of non-dipping of blood pressure at night was 62%. In our JingNing population study, we found that Chinese had a higher nighttime diastolic blood pressure than White populations, and the prevalence of isolated nocturnal hypertension was 10.9%. Patients with isolated nocturnal hypertension compared with normotensive subjects had an increased arterial stiffness. Thus, a preferable antihypertensive drug should not only reduce the 24-h mean level of blood pressure, but should also effectively control morning blood pressure surge and reduce nighttime blood pressure.

At present, there are two mechanisms of long-acting antihypertensive agents. One is that the compound itself has a long half life time and hence shows a long term effect. Another is that the efficacy of a short-acting drug is elongated by using a slow release or a controlled release (such as GITS) technique. However, the latter mechanism may vary between individuals because of the difference in the gastrointestinal function. Therefore, a long-acting compound should be more reliable in the maintenance of long term efficacy than slow release or controlled release agents. In the class of dihydropyridine calcium channel blockers, amlodipine is a long-acting compound because of a long half life time (up to 50 hours), and nifedipine GITS uses a controlled release technique. Several recent studies compared 24-h blood pressure lowering effect of these 2 drugs, but produced inconsistent results. At least one study suggested that amlodipine may prevent morning blood pressure rise more effectively than nifedipine GITS. However, other studies demonstrated similar effect on morning blood pressure control of these 2 drugs. The inconsistency might be attributable to a chance finding, because of the small sample size (less than 100). Therefore, a randomized controlled trial with a larger sample size is required to compare these 2 dihydropyridines in the blood pressure control over 24 hours in general and during early morning hours and at night in particular.

4. Objective: The primary objective of this study is to test the hypothesis that amlodipine compared with nifedipine GITS has a stronger effect in preventing morning blood pressure surge (4 am to 8 am) in mild to moderate hypertensive patients.

The secondary objective of the study is to compare the effects of amlodipine and nifedipine GITS in reducing nighttime blood pressure (10 pm to 4 am) in patients with a decreased nocturnal blood pressure fall.

5. Study design: The present study is designed as a randomized, actively controlled, multi-centre parallel group trial (phase Ⅳ) with two equally sized treatment groups: amlodipine and nifedipine GITS.

6. Study population: In 20 research-oriented university hospitals in China and in a pre-defined timeframe, 500 patients will be considered for inclusion into the present study according to the inclusion/exclusion criteria.

7. Randomization and treatment: After stratification for centre, 500 eligible patients will be randomized into 2 groups. 250 will receive amlodipine 5 mg per day, and 250 will receive nifedipine GITS 30 mg per day.

At 4 weeks of follow-up, the drug dosage per day may increase to 10 mg of amlodipine and 60 mg of nifedipine GITS, if blood pressure measured in doctor's office cannot be controlled to a level below 140/90 mm Hg. If there were no compelling indication, no other antihypertensive drug is allowed during the 2-month trial. All antihypertensive medication should be taken before breakfast from 6-8 clock in the morning.

8. Follow up: All patients should give written informed consent at entry into the present study. In addition to 24-h ambulatory blood pressure monitoring, patients should also undergo a questionnaire survey and clinical measurements including clinic blood pressure. Patients should be followed up in normal working hours in the morning or in the afternoon. The precise follow-up time of the day should be recorded. At each follow-up visit, the responsible physician should measure a patient's blood pressure and pulse rate, and collect information on the use of medications, serious adverse events, adverse events and cardiovascular complications. At 4 and 8 weeks of follow-up, 24-h and 48-h ambulatory blood pressure monitoring will be performed, respectively. When 48-h ambulatory blood pressure monitoring is performed at 8 weeks of follow-up, the patient should not take any antihypertensive medication on the second day of monitoring.

Only validated blood pressure monitors (SpaceLabs 90207 and 90217) will be used. Before each ambulatory blood pressure measurement, blood pressure monitors will be set up in a standardized way. A cuff of proper size should be secured to the left arm of the patient. Before the commencement of ambulatory blood pressure measurement, blood pressure will be measured twice using mercury sphygmomanometer. Immediately after these 2 measurements, blood pressure will be measured twice manually with the monitor. Then, blood pressure will be measured automatically according to predefined time intervals of the blood pressure monitor (every 20 minutes from 8 am to 10 pm and every 30 minutes from 10 pm to 8 am). At the end of ambulatory blood pressure monitoring, data will be transferred to a computer program. The same size cuff and the same arm should be used for all 3 ambulatory measurements for a patient. On the monitoring day, the patient should record the time to go to bed and to get up, the use of medications, and physical activity.

9. Potential difficulties: During the study, ambulatory blood pressure monitoring may fail because of less than 20 readings during the whole day, less than 10 readings in the daytime or less than 5 readings at night. These failed measurements will have to be repeated.

10. Sample size estimation and statistical analysis: It is projected that the standard deviation of morning blood pressure in the enrolled hypertensive patients is 12 mm Hg, and amlodipine, compared with nifedipine GITS, reduces morning blood pressure at 4 months of follow-up by 4 mm Hg. If α=0.05 and power=90%, the study will require a sample size of 190 hypertensive patients per group to detect the projected difference in the morning blood pressure (4 am-8 am). After accounting for 5% of drop out rate and 20% patients on add-on therapy, the sample size for each group is 250. Thus the number of required subject for the whole trial is 500.

The trial will mainly compare the amlodipine with nifedipine GITS group in the changes of morning blood pressure (4 am-8 am, about 8 blood pressure readings) and nighttime blood pressure (10 pm-4 am) at 4 and 8 weeks from baseline. The student t test will be used and 95% confidence interval of the differences between the 2 groups will be computed. In addition, an adjusted analysis (ANOVA) will also be performed while accounting for major baseline characteristics.

11. Timeline: The trial will start from October 2009, 500 eligible patients would be randomized and followed up for 2 months. Database construction and statistical analysis will take 3 months. The trial will be published at the international congresses and in the English and Chinese literature in 2013.

12. Organization: The principal investigator will be Professor Jiguang Wang from the Centre for Epidemiological Studies and Clinical Trials, Ruijin Hospital, Shanghai, China. Professor Yan Li from the same centre will be the coordinator of the trial. 20 research oriented hospitals will participate in the recruitment of the study subjects. At least 20 subjects should be recruited in each of the participating hospitals.

ELIGIBILITY:
Inclusion Criteria:

* Age: 40 to 70 years old.
* Untreated patients or those on monotherapy of antihypertensive drugs but with uncontrolled blood pressure in the ranges of 140-160/90-100 mmHg.
* Patients on antihypertensive medication should discontinue their antihypertensive treatment for at least 4 weeks. During the 4 weeks run-in period, all patients should have 2 clinic visits. At each visit, blood pressure will be measured 3 times consecutively. The average of these 6 readings from 2 clinic visits should be in the range of 140-180 systolic or 90-110 diastolic mm Hg. 24-h mean blood pressure should be equal to or higher than 130 mm Hg systolic and 80 mm Hg diastolic.
* The patients should sign the consent form prior to the participation in the trial, adhere to the study design, and can visit the outpatient clinic on his/her own.

Exclusion Criteria:

* With life-threatening disease.
* With myocardial infarction or stroke in the last 2 years.
* With contraindications to a dihydropyridine calcium channel blocker.
* Current participation in another trial or trials.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 510 (Actual)
Dates: Start 2009-10; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
the change from baseline in the mean systolic blood pressure during the morning hours (4 am to 8 am) of the first 24-hour ambulatory blood pressure monitoring at week 8 after randomization | 8 weeks

SECONDARY OUTCOMES:
the change from baseline in mean systolic blood pressure during the morning, mean systolic blood pressure at night, mean systolic blood pressure during the morning after missed dose, mean 24 h systolic blood pressure and mean daytime blood pressure | 4, 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jiguang Wang, MD, PhD, Principal Investigator — Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai Institite of Hypertension, Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, China